CLINICAL TRIAL: NCT00569569
Title: Retaane® in Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rudolf Foundation Clinic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFC012007
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Last update posted 2007-12-07 (Estimated); Status verified 2007-12

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients treated with Retaane
  Interventions: Drug: juxtascleral depot injection of Retaane

INTERVENTIONS:
Drug: juxtascleral depot injection of Retaane — juxtascleral depot injection of Retaane

SUMMARY:
The treatment of fibrotic choroidal neovascular lesions with presence of residual peripheral activity in age related macular degeneration currently presents a great challenge. With visual loss threatening, there are only very few therapeutic options.

While these patients are neither suitable for laser therapy nor for photodynamic therapy with Verteporfin, antiangiogenic drugs applied intravitreally are now available.

Some patients however reject this therapeutic option because of potential complications such as endophthalmitis and the frequency of necessary injections. 20 patients who rejected intravitreal therapy were treated with Anecortave acetate (Retaane®) which was applied as a juxtascleral depot injection.

ELIGIBILITY:
Inclusion Criteria:

* rejection of intravitreal injections
* presence of fibrotic choroidal neovascular lesions with presence of residual peripheral activity in age related macular degeneration

Exclusion Criteria:

* conditions precluding judgement of the fundus

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-02; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Increase in VA | 6 months

SECONDARY OUTCOMES:
Decrease in Macula Edema | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Binder, M.D., Study Chair — no affiliation